CLINICAL TRIAL: NCT00330772
Title: Pilot Study of Preoperative Aspirin and Postoperative Clopidogrel's Effects on Graft Patency and Cardiac Events in Coronary Artery Bypass Surgery
Brief Title: Preoperative Aspirin and Postoperative Antiplatelets in Coronary Artery Bypass Grafting: The PAPA CABG Study
Acronym: PAPA CABG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 06-091
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Grafting
Keywords: Cardiac Surger; Coronary Artery Bypass Grafting; Graft patency; Aspirin; Clopidogrel; Hemorrhage; Transfusion
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aspirin
Drug: Clopidogrel

SUMMARY:
Main Research Question(s):

What is the effect of continuing aspirin until the time of coronary artery bypass graft surgery and of adding clopidogrel to aspirin after coronary artery bypass graft surgery for preventing blockage of coronary grafts, heart attack, stroke, and death? To reliably answer this question requires a large randomised trial. Before applying for a major grant from the Canadian Institute for Health Research to do the large study we would like to perform a small pilot study of 150 patients to demonstrate that it is feasible to recruit patients and to use a new test called "CT angiography" to determine whether the bypass grafts are still working or have become blocked.

(ii) Why is this research important? Coronary artery bypass surgery has made a very important contribution to improving the health and survival of patients with advanced coronary artery disease but still has many problems. One in 10 patients experiences a heart attack at the time of surgery, 1 in 20 experiences a heart attack, stroke, or death during hospitalization, and 1 in 4 patients has at least 1 blocked graft within 1 year of surgery. Antiplatelet drugs such as aspirin and clopidogrel are effective for preventing heart attacks, strokes and deaths but aspirin is usually stopped before coronary artery bypass graft surgery because of concerns about increasing the risk of bleeding. The effectiveness of the combination of clopidogrel and aspirin after surgery has not been evaluated. Our pilot study will provide key information about feasibility that will help us to design and perform a large definitive study in the future.

(iii) What is being studied? We will be looking at blood flow in bypass grafts as well as the occurrence of heart attack, stroke, and death. For safety we will be looking at bleeding, transfusion, and need for further surgery because of bleeding. We will also perform laboratory tests of platelet function to measure and compare the effect of the study treatments to prevent blood clots from forming.

DETAILED DESCRIPTION:
BACKGROUND: Platelets play a central role in the pathogenesis of ischemic complications (coronary artery bypass graft occlusion, myocardial infarction, stroke) following CABG surgery. Aspirin and clopidogrel used alone or in combination are effective for preventing ischemic complications in a broad range of high risk patients. However aspirin is usually discontinued before CABG surgery because of concerns about bleeding while the combination of aspirin and clopidogrel has not been evaluated for preventing ischemic complications after CABG surgery.

OBJECTIVES: The overall objectives of our research are to compare the effectiveness and safety of aspirin vs placebo before bypass surgery, and clopidogrel plus aspirin vs aspirin alone after surgery, on:

1. blockage of coronary artery bypass grafts, MI, stroke, or death at 30 days
2. bleeding and need for transfusion after surgery The specific objective of the present pilot study is to demonstrate the feasibility of recruiting patients undergoing CABG surgery into this study and of performing CT angiography at 30 days to determine graft patency. We will also measure the effect of different antiplatelet treatments on platelet function and blood markers of systemic inflammation during the first 48 hours after surgery.

DESIGN: This is a 2x2 factorial study of 150 elective CABG patients who will be randomized to receive low dose aspirin (81mg/d) or placebo for 5 days prior to surgery and aspirin 325mg loading dose followed by 81 mg/d plus clopidogrel 75 mg/d versus aspirin 81 mg/d and placebo post operatively.

OUTCOME: graft patency measured by CT angiography, MI, stroke, death, bleeding, transfusion requirement, need for re-exploration surgery, and laboratory measures of platelet function and aspirin resistance (including 11-dehydro thromboxane B2).

SAMPLE SIZE: This is a pilot study designed primarily to demonstrate feasibility. We propose to recruit a total of 150 patients over a 12 month period (2-4 per week).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Undergoing on-pump, elective coronary artery bypass grafting with at least 2 free grafts
* Patient able to give informed consent

Exclusion Criteria:

* planned date of surgery is <5 days from planned recruitment date
* patient has clear indication for anticoagulation (eg. mechanical heart valve, atrial fibrillation) or ADP receptor antagonist (eg. drug-eluting stent)
* allergy to or intolerance of aspirin or clopidogrel
* history of bleeding diathesis, significant GI bleed, ICH, or liver failure
* Patient has known renal failure or contraindication for Cardiac CT Angio
* Patient has had previous cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Graft patency, MI, Death, Stroke

SECONDARY OUTCOMES:
Bleeding, transfusion, re-exploration, Platelet function tests

CONTACTS AND LOCATIONS:
Overall Officials: Jack CJ Sun, MD, Principal Investigator — McMaster University; John W Eikelboom, MD, MSc, Study Director — McMaster University; Kevin HT Teoh, MD, Study Chair — McMaster University; Salim Yusuf, MD, DPhil, Study Chair — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Sun JC, Teoh KH, Lamy A, Sheth T, Ellins ML, Jung H, Yusuf S, Anand S, Connolly S, Whitlock RP, Eikelboom JW. Randomized trial of aspirin and clopidogrel versus aspirin alone for the prevention of coronary artery bypass graft occlusion: the Preoperative Aspirin and Postoperative Antiplatelets in Coronary Artery Bypass Grafting study. Am Heart J. 2010 Dec;160(6):1178-84. doi: 10.1016/j.ahj.2010.07.035. PMID 21146675